CLINICAL TRIAL: NCT03025815
Title: Effects of the Oral Stimulation Program in Extreme Preterm Infants: A Randomized Clinical Trial
Brief Title: Effects of the Oral Stimulation Program in Extreme Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 41366915.5.0000.5327
Record Dates: First submitted 2017-01-02; First posted 2017-01-20 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Infant, Premature; Feeding Behavior
Keywords: Infant, Premature
MeSH Terms: conditions — Premature Birth; Feeding Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Oral stimulation program consists of the a 15 minutes stimulation program, whereby the first 12 minutes involved stroking the cheeks, lips, gums, and tongue, and the final 3 minutes consists of sucking on a pacifier routinely.
  Interventions: Other: Intervention group
- Control group (Sham Comparator): sham stimulation program consists of the same researcher placing her hands for 15 minutes.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — Oral stimulation program consists of the a 15 minutes stimulation program, whereby the first 12 minutes involved stroking the cheeks, lips, gums, and tongue, and the final 3 minutes consists of sucking on a pacifier routinely.
  Other Names: Oral stimulation program
  Arms: Intervention group
Other: Control group — sham stimulation program consists of the same researcher placing her hands for 15 minutes.
  Other Names: Sham stimulation program
  Arms: Control group

SUMMARY:
The purpose of this study is to determine whether oral stimulation program are effective to improve oral feeding efficiency. The sample size estimated in 74 preterm, randomized classification of the subjects into to experimental and a control group.

DETAILED DESCRIPTION:
Recent studies have suggested that an oral stimulation program applied to preterm infants facilitates their oral feeding progress, improve breastfeeding rates in preterm infants and decreases the length of hospital stay. The objective of this study will evaluate the effect an oral stimulation program on the performance feeding, the length of the transition oral feeding, length of hospital stay and breastfeeding rates upon discharge.

Primarily, will be evaluated the effect an oral stimulation program on the performance feeding. All infants will be assessed by a speech pathologist blinded as to the group randomization.

Secondarily, will be observed the length of the transition oral feeding of the preterm infants, conducted by medical team and will be observed length of hospital stay. Both groups will be monitored from when they were assigned to participate in the study until hospital discharge.

All statistical will be conducted using Statistical Package for Social Sciences® version 18.0. The data will be analyzed for treatment group differences with chi-square or Fisher's exact tests for the categorical variables and with non-parametric tests for the continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* infants with between 26 and 32 weeks gestational age as determined by date of last menstruation and first trimester ultrasound or by clinical examination.

Exclusion Criteria:

* infants with medical complications, such as grades III or IV intraventricular hemorrhage or periventricular leukomalacia
* congenital diseases such as chromosomal or genetic abnormalities
* bronchopulmonary dysplasia
* necrotizing enterocolitis.

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Oral feeding performance | 20 minutes
  The volume transfer is as considered as the percentage of the volume consumed (%).

SECONDARY OUTCOMES:
Oral feeding transition time | 60 days
  number of days
Days hospital stay | 6 months
  number of days

CONTACTS AND LOCATIONS:
Overall Officials: Rita C Silveira, Professor, Principal Investigator — Neonatal Section
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] da Rosa Pereira K, Levy DS, Procianoy RS, Silveira RC. Impact of a pre-feeding oral stimulation program on first feed attempt in preterm infants: Double-blind controlled clinical trial. PLoS One. 2020 Sep 9;15(9):e0237915. doi: 10.1371/journal.pone.0237915. eCollection 2020. PMID 32903261